CLINICAL TRIAL: NCT03941600
Title: Feasibility of a Community-based Exercise Intervention for Persons With Spinal Cord Injury
Brief Title: Feasibility of Exercise and Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kerri Morgan, Assistant Professor of Occupational Therapy and Neurology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201809174; K12HD055931 (NIH)
Record Dates: First submitted 2019-01-18; First posted 2019-05-08 (Actual); Results first posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-01

CONDITIONS: Spinal Cord Injuries
Keywords: occupational therapy; exercise
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community-based Exercise Intervention group (CBEI) (Active Comparator): A group performing a 12-week guided exercise program at an accessible community health and wellness center
  Interventions: Behavioral: Community-based Exercise Intervention group (CBE)
- Exercise Education Control group (EEG) (Placebo Comparator): A group receiving educational information about physical activity and exercise at home and then self-direction a 12-week exercise program on their own.
  Interventions: Behavioral: Exercise Education Control group (EEG)

INTERVENTIONS:
Behavioral: Community-based Exercise Intervention group (CBE) — The CBEI group will receive 36 (60-90 minute) one-on-one, formally directed exercise sessions by trained staff over 12 weeks. By the end the goal is to have the participants guiding their own regimens. Personalized sessions will be created for each participant based on their fitness goal(s) and preferences. Each session will include vitals, pain assessment, warm-up, stretching, cardiovascular, and strength exercises and cool-down. The participants will be monitored to ensure they are achieving at least 30 minutes of moderate-to-vigorous exercise 3 times a week. Activity monitors will also be worn to capture intensity data. At the end of each session, participants will describe their likes and dislike as well as what they gained and what they suggest for improvement. At the end of each session, the trainer will rate the participant's perceived participation during the session (1-6) using the Pittsburgh Rehabilitation Participation Scale.
  Arms: Community-based Exercise Intervention group (CBEI)
Behavioral: Exercise Education Control group (EEG) — The EEG group will complete an intervention that consists of a one-on-one, hour-long educational session orienting participants to an online resource center, the National Center on Health, Physical Activity, and Disability (NCHPAD). NCHPAD promotes health and well-being for PwD through resources such as adapted exercise videos, information on accessible fitness equipment, personalized exercise videos tailored to PwD, and an individualized 14-week exercise program. Participants will be given an overview of NCHPAD and asked to identify resources of interest on the website. Each participant will be asked to use resources on NCHPAD to engage in physical activity for 12 weeks. Each participant will receive a weekly phone call to inquire about their physical activity, exercises engaged in, RPE during exercise, and whether any resources were used.
  Arms: Exercise Education Control group (EEG)

SUMMARY:
The purpose of the study is to examine the impact of a community-based exercise intervention (CBEI) for persons with spinal cord injury (PwSCI) on physiological and psychological well-being and identify barriers and facilitators to implementation.

DETAILED DESCRIPTION:
People with spinal cord injury (PwSCI) are at a greater risk for major health conditions and poorer health outcomes than the population without spinal cord injury. For PwSCI, habitual exercise is critical for both physiological and psychological well-being. Prior research indicates that exercise programs conducted in a controlled setting have positive effects on the physical and psychosocial fitness of PwSCI, but the efficacy and feasibility of these programs are not well understood in community-based settings. The proposed project aims to examine potential health benefits in response to the intervention and identify the barriers and facilitators to successful implementation of a CBEI in PwSCI. The long-term goal of this research is to improve health outcomes of PwSCI by identifying strategies to promote health and support exercise in the community.

The project research aims are to:

1. Estimate improvements in physical function, cardio-metabolic health, and psychological well-being of participants enrolled in a CBEI compared to an education-only group.
2. Identify barriers, facilitators, and reasons for positive determinants for PwSCI to exercise in a community-based setting.

A single-blind pilot RCT will be conducted. Forty individuals with SCI will be recruited. Each participant will be randomized into either a 12-week CBEI (n=20) or an education control group (n=20). Participants' cardiorespiratory fitness, body composition, metabolic blood chemistries and strength will be assessed pre- (T1) and post- (T2) intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SCI
* 18 years or older
* Have written physician approval to participate in the study
* Ability to use upper extremities to exercise
* Participate in < 60 minutes of moderate-intensity exercise per week in the last month
* Understand English at a sixth-grade level or higher
* Be able to follow multi-step instructions
* Independently provide informed consent
* Willing to participate in three assessments and 36 intervention sessions

Exclusion Criteria:

* Enrollment in a structured exercise program in the past six months.
* Have had cardiovascular complications within the past year
* Currently receive medical treatment for an acute upper extremity injury
* Have a Stage IV pressure injury
* Have a cognitive impairment that does not allow them to provide consent or follow multi-step directions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerri A Morgan, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] National Spinal Cord Injury Statistical Center. (2016). 2016 Annual Statistical Report - Complete Public Version. Birmingham, AL: University of Alabama at Birmingham.
- [Background] Keyser RE, Rasch EK, Finley M, Rodgers MM. Improved upper-body endurance following a 12-week home exercise program for manual wheelchair users. J Rehabil Res Dev. 2003 Nov-Dec;40(6):501-10. doi: 10.1682/jrrd.2003.11.0501. PMID 15077662
- [Background] West CR, Alyahya A, Laher I, Krassioukov A. Peripheral vascular function in spinal cord injury: a systematic review. Spinal Cord. 2013 Jan;51(1):10-9. doi: 10.1038/sc.2012.136. Epub 2012 Nov 27. PMID 23184028
- [Background] Froehlich-Grobe K, Jones D, Businelle MS, Kendzor DE, Balasubramanian BA. Impact of disability and chronic conditions on health. Disabil Health J. 2016 Oct;9(4):600-8. doi: 10.1016/j.dhjo.2016.04.007. Epub 2016 May 3. PMID 27216441
- [Background] Nightingale TE, Metcalfe RS, Vollaard NB, Bilzon JL. Exercise Guidelines to Promote Cardiometabolic Health in Spinal Cord Injured Humans: Time to Raise the Intensity? Arch Phys Med Rehabil. 2017 Aug;98(8):1693-1704. doi: 10.1016/j.apmr.2016.12.008. Epub 2017 Jan 13. PMID 28089898
- [Background] Hicks AL, Martin Ginis KA, Pelletier CA, Ditor DS, Foulon B, Wolfe DL. The effects of exercise training on physical capacity, strength, body composition and functional performance among adults with spinal cord injury: a systematic review. Spinal Cord. 2011 Nov;49(11):1103-27. doi: 10.1038/sc.2011.62. Epub 2011 Jun 7. PMID 21647163
- [Background] Carroll DD, Courtney-Long EA, Stevens AC, Sloan ML, Lullo C, Visser SN, Fox MH, Armour BS, Campbell VA, Brown DR, Dorn JM; Centers for Disease Control and Prevention (CDC). Vital signs: disability and physical activity--United States, 2009-2012. MMWR Morb Mortal Wkly Rep. 2014 May 9;63(18):407-13. PMID 24807240
- [Background] Ginis KA, Arbour-Nicitopoulos KP, Latimer AE, Buchholz AC, Bray SR, Craven BC, Hayes KC, Hicks AL, McColl MA, Potter PJ, Smith K, Wolfe DL. Leisure time physical activity in a population-based sample of people with spinal cord injury part II: activity types, intensities, and durations. Arch Phys Med Rehabil. 2010 May;91(5):729-33. doi: 10.1016/j.apmr.2009.12.028. PMID 20434610
- [Background] Sullivan KJ. President's perspectives. Healthcare Reform: a call to action for our patients. J Neurol Phys Ther. 2009 Sep;33(3):171-2. doi: 10.1097/NPT.0b013e3181b65372. No abstract available. PMID 19809396
- [Background] McCormick ZL, Lynch M, Liem B, Jacobs G, Hwang P, Hornby TG, Rydberg L, Roth E. Feasibility for developing cardiovascular exercise recommendations for persons with motor-complete paraplegia based on manual wheelchair propulsion; A protocol and preliminary data. J Spinal Cord Med. 2016;39(1):45-9. doi: 10.1179/2045772314Y.0000000292. Epub 2015 Jan 13. PMID 25582138
- [Background] Kaye, H. S., Kang, T., & LaPlante, M. P. (2000). Mobility device use in the United States. (No. 14). Washington, DC: U.S. Department of Education, National Institute on Disability and Rehabilitation Research.
- [Background] Zwinkels M, Verschuren O, Janssen TW, Ketelaar M, Takken T; Sport-2-Stay-Fit study group; Sport-2-Stay-Fit study group. Exercise training programs to improve hand rim wheelchair propulsion capacity: a systematic review. Clin Rehabil. 2014 Sep;28(9):847-61. doi: 10.1177/0269215514525181. Epub 2014 Mar 10. PMID 24615862
- [Background] American College of Sports Medicine. (2014). ACSM's Guidelines for Exercise Testing and Prescription (9th ed.). Philadelphia: Lippincott Williams & Wilkins.
- [Background] Totosy de Zepetnek JO, Pelletier CA, Hicks AL, MacDonald MJ. Following the Physical Activity Guidelines for Adults With Spinal Cord Injury for 16 Weeks Does Not Improve Vascular Health: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2015 Sep;96(9):1566-75. doi: 10.1016/j.apmr.2015.05.019. Epub 2015 Jun 10. PMID 26070976
- [Background] Gebel K, Ding D, Chey T, Stamatakis E, Brown WJ, Bauman AE. Effect of Moderate to Vigorous Physical Activity on All-Cause Mortality in Middle-aged and Older Australians. JAMA Intern Med. 2015 Jun;175(6):970-7. doi: 10.1001/jamainternmed.2015.0541. PMID 25844882
- [Background] Weston KS, Wisloff U, Coombes JS. High-intensity interval training in patients with lifestyle-induced cardiometabolic disease: a systematic review and meta-analysis. Br J Sports Med. 2014 Aug;48(16):1227-34. doi: 10.1136/bjsports-2013-092576. Epub 2013 Oct 21. PMID 24144531
- [Background] Ramos JS, Dalleck LC, Tjonna AE, Beetham KS, Coombes JS. The impact of high-intensity interval training versus moderate-intensity continuous training on vascular function: a systematic review and meta-analysis. Sports Med. 2015 May;45(5):679-92. doi: 10.1007/s40279-015-0321-z. PMID 25771785
- [Background] Jelleyman C, Yates T, O'Donovan G, Gray LJ, King JA, Khunti K, Davies MJ. The effects of high-intensity interval training on glucose regulation and insulin resistance: a meta-analysis. Obes Rev. 2015 Nov;16(11):942-61. doi: 10.1111/obr.12317. PMID 26481101
- [Background] Yim SY, Cho KJ, Park CI, Yoon TS, Han DY, Kim SK, Lee HL. Effect of wheelchair ergometer training on spinal cord-injured paraplegics. Yonsei Med J. 1993 Sep;34(3):278-86. doi: 10.3349/ymj.1993.34.3.278. PMID 8259705
- [Background] Klaesner J, Morgan KA, Gray DB. The development of an instrumented wheelchair propulsion testing and training device. Assist Technol. 2014 Spring;26(1):24-32. doi: 10.1080/10400435.2013.792020. PMID 24800451
- [Background] U.S. Department of Health and Human Services (2008). 2008 Physical Activity Guidelines for Americans. Washington, D. C.: U.S. Department of Health and Human Services.
- [Background] Stinson JN, Kavanagh T, Yamada J, Gill N, Stevens B. Systematic review of the psychometric properties, interpretability and feasibility of self-report pain intensity measures for use in clinical trials in children and adolescents. Pain. 2006 Nov;125(1-2):143-57. doi: 10.1016/j.pain.2006.05.006. Epub 2006 Jun 13. PMID 16777328
- [Background] Gray DB, Hollingsworth HH, Stark SL, Morgan KA. Participation survey/mobility: psychometric properties of a measure of participation for people with mobility impairments and limitations. Arch Phys Med Rehabil. 2006 Feb;87(2):189-97. doi: 10.1016/j.apmr.2005.09.014. PMID 16442971
- [Background] Cowan RE, Callahan MK, Nash MS. The 6-min push test is reliable and predicts low fitness in spinal cord injury. Med Sci Sports Exerc. 2012 Oct;44(10):1993-2000. doi: 10.1249/MSS.0b013e31825cb3b6. PMID 22617394
- [Background] Heymsfield SB, Smith R, Aulet M, Bensen B, Lichtman S, Wang J, Pierson RN Jr. Appendicular skeletal muscle mass: measurement by dual-photon absorptiometry. Am J Clin Nutr. 1990 Aug;52(2):214-8. doi: 10.1093/ajcn/52.2.214. PMID 2375286
- [Background] Damirchi A, Tehrani BS, Alamdari KA, Babaei P. Influence of aerobic training and detraining on serum BDNF, insulin resistance, and metabolic risk factors in middle-aged men diagnosed with metabolic syndrome. Clin J Sport Med. 2014 Nov;24(6):513-8. doi: 10.1097/JSM.0000000000000082. PMID 24662570
- [Background] Berg U, Bang P. Exercise and circulating insulin-like growth factor I. Horm Res. 2004;62 Suppl 1:50-8. doi: 10.1159/000080759. PMID 15761233
- [Background] Fabel K, Fabel K, Tam B, Kaufer D, Baiker A, Simmons N, Kuo CJ, Palmer TD. VEGF is necessary for exercise-induced adult hippocampal neurogenesis. Eur J Neurosci. 2003 Nov;18(10):2803-12. doi: 10.1111/j.1460-9568.2003.03041.x. PMID 14656329
- [Background] Kroll T, Barbour R, Harris J. Using focus groups in disability research. Qual Health Res. 2007 May;17(5):690-8. doi: 10.1177/1049732307301488. PMID 17478650
- [Background] Krueger, R. A. & Casey, M. A. (2009). Focus Groups: A Practical Guide for Applied Research (4th ed.). Thousand Oaks, CA: Sage.
- [Background] Bailey RR, Klaesner JW, Lang CE. An accelerometry-based methodology for assessment of real-world bilateral upper extremity activity. PLoS One. 2014 Jul 28;9(7):e103135. doi: 10.1371/journal.pone.0103135. eCollection 2014. PMID 25068258
- [Background] Garcia-Masso X, Serra-Ano P, Garcia-Raffi LM, Sanchez-Perez EA, Lopez-Pascual J, Gonzalez LM. Validation of the use of Actigraph GT3X accelerometers to estimate energy expenditure in full time manual wheelchair users with spinal cord injury. Spinal Cord. 2013 Dec;51(12):898-903. doi: 10.1038/sc.2013.85. Epub 2013 Sep 3. PMID 23999111
- [Background] Morgan, K. A., Engsberg, J. R., & Klaesner, J. (2015). The testing of an instrumented wheelchair propulsion testing and training device. Journal of Physical Medicine, Rehabilitation and Disabilities, 1(003), 1-9.
- [Background] Evans N, Wingo B, Sasso E, Hicks A, Gorgey AS, Harness E. Exercise Recommendations and Considerations for Persons With Spinal Cord Injury. Arch Phys Med Rehabil. 2015 Sep;96(9):1749-50. doi: 10.1016/j.apmr.2015.02.005. Epub 2015 Jul 18. No abstract available. PMID 26198424

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Community-based Exercise Intervention Group (CBEI) | Exercise Education Control Group (EEG)
Started | 27 | 22
Completed | 15 | 17
Not Completed | 12 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Community-based Exercise Intervention Group (CBEI) | Exercise Education Control Group (EEG) | Total
Number analyzed (Participants) | 27 | 22 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.04 (10.847) | 40.77 (15.991) | 39.27 (13.323)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 20 | 17 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 11 | 27
  White | 7 | 8 | 15
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 27 | 22 | 49

OUTCOME MEASURES:

1. Primary Outcome: VO2 Peak - Cardiorespiratory Fitness Change (Peak Oxygen Consumption Change)
Description: VO2 peak will be measured using a standard computer-integrated, open-circuit, breath-by-breath metabolic measurement system (TrueOne 2400, Parvo Medics, Sandy UT) while the participant performs a graded-exercise test on an arm crank ergometer (SCIFIT PRO2, Life Fitness, Tulsa, OK). The protocol involves a 3-minute warm-up followed by a standard ramp protocol which is typically completed in 8-12 minutes.
Time Frame: Baseline and Up to 4 weeks post intervention
Population: Only valid data was analyzed. Data deemed "valid" when the following criteria was met, (before/within 1 minute of cooldown, RER =/> 1.1, RPE reported as =/>15. A participant's PRE/POST scores both had to be valid to be included in analysis. CBEI group = 6 participants excluded, 3 did not have any valid VO2 test, 3 only had 1 valid VO2 test. EEG group = 1 did not have any valid VO2 test, 2 only had 1 valid VO2 test, 1 participant was unable to physically complete the test.
Measure: Mean (Standard Error); unit: ml/kg/min
Arm/Group | Community-based Exercise Intervention Group (CBEI) | Exercise Education Control Group (EEG)
Number analyzed (Participants) | 9 | 13
ml/kg/min
  Pre | 14.69 (1.22) | 14.36 (1.28)
  Post | 15.61 (1.95) | 13.74 (1.09)

2. Primary Outcome: DEXA - Body Composition Overall Body Fat % Change
Description: Participants will then undergo body composition assessment via DEXA (General Electric Lunar iDXA), which is commonly used in research due to its precision and safety. Body fat % will be the unit of measure.
Time Frame: Baseline and Up to 4 weeks post intervention
Population: Only 2 participants (both from the CBEI group) were able to complete this outcome measure due to the COVID-19 pandemic. Our research project was considered non-essential and therefore the services to conduct these assessments were shut down and not available.
Measure: Mean (Standard Error); unit: percentage of body fat
Arm/Group | Community-based Exercise Intervention Group (CBEI) | Exercise Education Control Group (EEG)
Number analyzed (Participants) | 2 | 0
percentage of body fat
  Pre | 39.800 (.1000) |
  Post | 38.750 (2.2500) |

3. Primary Outcome: Metabolic Blood Chemistries - HbA1c Level Change
Description: Blood draws will be completed to measure HbA1c levels in %. Participants will fast 8-10 hours prior to blood draw.
Time Frame: Baseline and Up to 4 weeks post intervention
Population: This data was only collected on 2 participants (1 CBEI group and 1 EEG group) at the pre-assessment period and 3 participants (2 CBEI group and 1 EEG group) at post assessment. We were not able to complete this outcome measure on any further participants due to the COVID-19 pandemic. Our research project was considered non-essential and therefore the services to conduct these assessments were shut down and not available.
Measure: Mean (Standard Error); unit: percentage of HbA1c levels
Arm/Group | Community-based Exercise Intervention Group (CBEI) | Exercise Education Control Group (EEG)
Number analyzed (Participants) | 2 | 1
percentage of HbA1c levels
  Pre: number analyzed (Participants) | 1 | 1
  Pre | 4.9 | 5.0
  Post | 4.9 (.4000) | 5.0

4. Primary Outcome: Metabolic Blood Chemistries - Cholesterol Change
Description: Blood draws will be completed to measure cholesterol levels. Unit of measure will be in mg/dL. Participants will fast 8-10 hours prior to blood draw.
Time Frame: Baseline and Up to 4 weeks post interventions
Population: Only 3 participants (2 CBEI and 1 EEG) were able to complete this outcome measure due to the COVID-19 pandemic. Our research project was considered non-essential and therefore the services to conduct these assessments were shut down and not available.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Community-based Exercise Intervention Group (CBEI) | Exercise Education Control Group (EEG)
Number analyzed (Participants) | 2 | 1
mg/dL
  Pre | 172 (39) | 188
  Post | 170. (50) | 212

5. Secondary Outcome: Upper Extremity Strength - Upper Body Strength Change
Description: Strength will be measured via isotonic 1RM testing unilaterally on four upper-extremity exercises (chest press, back row, rickshaw, biceps flexion) using a BTE™ PrimusRS (BTE™, Hanover, MD). Data was organized into one single strength variable by summing the 4 left side upper extremity exercises together, then summing the 4 right side upper extremity exercises together, and finally taking those 2 totals (from left side and right side) and summing them into one strength variable. A higher number indicates more strength. The BTE™ PrimusRS uses an inch-pound (the torque of one pound of force applied to one inch of distance from the pivot) as it's unit of measurement.
Time Frame: Baseline and Up to 4 weeks post intervention
Population: 1 participant from the Excercise Education Control group (EEG) was unable to do the PRE upper extremity strength measure at baseline.
Measure: Mean (Standard Error); unit: inch-pound
Arm/Group | Community-based Exercise Intervention Group (CBEI) | Exercise Education Control Group (EEG)
Number analyzed (Participants) | 15 | 17
inch-pound
  Pre: number analyzed (Participants) | 15 | 16
  Pre | 287.83 (29.87) | 277.0 (28.17)
  Post | 351.37 (31.89) | 315.47 (29.44)

6. Secondary Outcome: PROMIS - Fatigue Short Form 8a
Description: Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue - assesses a range of self-reported fatigue symptoms over the past 7 days. PROMIS instruments are scored using item-level calibrations. Each question is answered using a 5-point Likert scale from "not at all (1)" to "very much (5)" with a raw score between 8 and 40. The t-score was automatically calculated using REDCap auto-score. A t-score of 50 indicates the mean score for the general population with a standard deviation of 10. A higher score reflects more of the domain being assessed. A t-score of 55-60 indicates mild fatigue, a t-score of 60-70 indicates moderate fatigue and a t-score of 70 or above indicates severe fatigue.
Time Frame: Baseline and Up to 4 weeks post intervention
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Community-based Exercise Intervention Group (CBEI) | Exercise Education Control Group (EEG)
Number analyzed (Participants) | 15 | 17
T-score
  Pre | 48.09 (1.49) | 49.31 (2.53)
  Post | 46.71 (1.66) | 50.43 (1.73)

7. Secondary Outcome: PROMIS - Emotional Distress - Depression - Short Form 8a
Description: Patient Reported Outcomes Measurement Information System (PROMIS) Emotional distress - Depression - assesses self-reported negative mood, views of self, social cognition, as well as decreased positive affect and engagement over the past 7 days. PROMIS instruments are scored using item-level calibrations. Each question is answered using a 5-point Likert scale from "never (1)" to "always (5)" with a raw score between 8 and 40. The t-score was automatically calculated using REDCap auto-score. A t-score of 50 indicates the mean score for the general population with a standard deviation of 10. A higher score reflects more of the domain being assessed. A t-score of 55-60 indicates mild depression, a t-score of 60-70 indicates moderate depression and a t-score of 70 or above indicates severe depression.
Time Frame: Baseline and Up to 4 weeks post intervention
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Community-based Exercise Intervention Group (CBEI) | Exercise Education Control Group (EEG)
Number analyzed (Participants) | 15 | 17
T-score
  Pre | 47.21 (2.36) | 51.44 (2.92)
  Post | 45.31 (1.75) | 51.69 (2.48)

8. Secondary Outcome: PROMIS - Pain Intensity - Short Form 3a
Description: Patient Reported Outcomes Measurement Information System (PROMIS) Pain Intensity - assesses how much a person hurts over the past 7 days. PROMIS instruments are scored using item-level calibrations. Each question is answered using a 5-point Likert scale from "had no pain (1)" to "very severe (5)" with a raw score between 3 and 15. The t-score was automatically calculated using REDCap auto-score. A t-score of 50 indicates the mean score for the general population with a standard deviation of 10. A higher score reflects more of the domain being assessed. A t-score of 55-60 indicates mild pain intensity, a t-score of 60-70 indicates moderate pain intensity and a t-score of 70 or above indicates severe pain intensity.
Time Frame: Baseline and Up to 4 weeks post intervention
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Community-based Exercise Intervention Group (CBEI) | Exercise Education Control Group (EEG)
Number analyzed (Participants) | 15 | 17
T-score
  Pre | 46.23 (3.37) | 45.08 (2.10)
  Post | 45.01 (3.23) | 45.43 (2.52)

9. Secondary Outcome: PROMIS - Pain Interference - Short Form 8a
Description: Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference - assesses self-reported consequences of pain on relevant aspects of one's life over the past 7 days, this includes how pain hinders engagement with social, cognitive, emotional, physical and recreational activities. PROMIS instruments are scored using item-level calibrations. Each question is answered using a 5-point Likert scale from "not at all (1)" to "very much (5)" with a raw score between 8 and 40. The t-score was automatically calculated using REDCap auto-score. A t-score of 50 indicates the mean score for the general population with a standard deviation of 10. A higher score reflects more of the domain being assessed. A t-score of 55-60 indicates mild pain interference, a t-score of 60-70 indicates moderate pain interference and a t-score of 70 or above indicates severe pain interference.
Time Frame: Baseline and Up to 4 weeks post intervention
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Community-based Exercise Intervention Group (CBEI) | Exercise Education Control Group (EEG)
Number analyzed (Participants) | 15 | 17
T-score
  Pre | 52.24 (2.6) | 52.06 (2.51)
  Post | 52.64 (2.64) | 51.96 (2.17)

10. Secondary Outcome: PROMIS - Sleep Disturbance - Short Form 8a
Description: Patient Reported Outcomes Measurement Information System (PROMIS) Sleep - assesses self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep over the past 7 days. PROMIS instruments are scored using item-level calibrations. Each question is answered using a 5-point Likert scale from "very poor (1)" to "very good (5)" with a raw score between 8 and 40. The t-score was automatically calculated using REDCap auto-score. A t-score of 50 indicates the mean score for the general population with a standard deviation of 10. A higher score reflects more of the domain being assessed. A t-score of 55-60 indicates mild sleep disturbance, a t-score of 60-70 indicates moderate sleep disturbance and a t-score of 70 or above indicates severe sleep disturbance.
Time Frame: Baseline and Up to 4 weeks post intervention
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Community-based Exercise Intervention Group (CBEI) | Exercise Education Control Group (EEG)
Number analyzed (Participants) | 15 | 17
T-score
  Pre | 48.71 (2.36) | 50.48 (2.63)
  Post | 48.87 (3.49) | 51.31 (2.77)

11. Secondary Outcome: PROMIS - Emotional Support
Description: Patient Reported Outcomes Measurement Information System (PROMIS) Emotional Support - assesses perceived feelings of being cared for and valued as a person and having confident relationships. PROMIS instruments are scored using item-level calibrations. Each question is answered using a 5-point Likert scale from "never (1)" to "always (5)". The t-score was automatically calculated using REDCap auto-score. A t-score of 50 indicates the mean score for the general population with a standard deviation of 10. A higher score reflects more of the domain being assessed. A t-score of 40-60 indicates an average amount of emotional support, a t-score of 60-70 indicates high levels of emotional support, and a t-score of 70 or above indicates very high levels of emotional support.
Time Frame: Baseline and Up to 4 weeks post intervention
Population: One participant within the Community-based Exercise Intervention group (CBEI) post data was missing, therefore only 14 were analyzed instead of 15
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Community-based Exercise Intervention Group (CBEI) | Exercise Education Control Group (EEG)
Number analyzed (Participants) | 15 | 17
T-score
  Pre | 55.77 (2.47) | 49.66 (1.94)
  Post: number analyzed (Participants) | 14 | 17
  Post | 55.01 (2.39) | 49.58 (1.63)

ADVERSE EVENTS:
Time Frame: We collected adverse event data for approximately 6 months on each individual and tracked adverse events on all participants through the entirety of the study.
Arm/Group | Community-based Exercise Intervention Group (CBEI) | Exercise Education Control Group (EEG)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/22
Other Adverse Events (participants affected / at risk) | 0/27 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT03941600/Prot_SAP_000.pdf